CLINICAL TRIAL: NCT00315185
Title: Phase II Study as First Line Treatment for Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Study of Paclitaxel, Carboplatin, and Cetuximab for Advanced Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPN-TH-017
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Last update posted 2010-09-23 (Estimated); Status verified 2010-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Advanced Non-small Cell Lung Cancer; First Line Treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Cetuximab

SUMMARY:
The purpose of this study is to determine the role of cetuximab (Erbitux) with chemotherapy for advanced colorectal carcinoma. This study will determine if this new agent can improve one's response to standard treatment.

DETAILED DESCRIPTION:
This research study is being done to determine if cetuximab will improve efficacy of standard chemotherapy. This agent targets epidermal growth factor receptor (EGFR). EGFR sits on the outside of tumor cells and controls tumor cell growth. This agent has been looked at alone and with other chemotherapy drugs in non-small-cell lung cancer (NSCLC). It has shown to be safe and can shrink tumors. There is little information about the combination of this agent with both paclitaxel and carboplatin. This study combines cetuximab with monthly carboplatin and weekly paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented stage IIIB or IV NSCLC
* Measurable disease
* ECOG performance status of 0-1
* Asymptomatic brain metastasis; must have completed radiotherapy/radiosurgery at least 2 weeks prior to enrollment and be off steroids.
* Radiotherapy must have been completed > 2 weeks prior to enrollment and patients must have recovered from adverse events of radiotherapy.
* >/= 18 years of age
* Adequate hematologic function: absolute neutrophil count (ANC) >/= 1,500/mm3; platelets >/= 100,000/mm3.
* Adequate hepatic function: total bilirubin </= 1.5 X upper limit of normal (ULN); AST and ALT </= 2.5 X ULN.
* Adequate renal function: serum creatinine </= 1.5mg/dL or creatinine clearance >/= 50cc/minute if serum creatinine > 1.5
* Signed an approved informed consent for this protocol and an approved informed consent for Health Insurance Portability and Accountability Act (HIPAA)
* EGFR status by immunohistochemistry (IHC) if sufficient tissue is available

Exclusion Criteria:

* Women of childbearing potential who have a positive pregnancy test at enrollment or within 7 days of treatment. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth regulation/control. Note: Patients are considered to not be of childbearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.
* Patients who have had prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for 3 years.
* Patients with significant history of cardiac disease, i.e., uncontrolled hypertension, unstable angina, uncontrolled congestive heart failure, myocardial infarction within the past year, cardiomyopathy with decreased ejection fraction, or cardiac ventricular arrythmias within the last year requiring new treatment .
* Patients with an uncontrolled seizure disorder, or active neurological disease.
* Patients with symptomatic brain metastasis.
* Patients who have received prior systemic chemotherapy.
* Patients who have received prior cetuximab or other therapy which specifically and directly targets the EGF pathway.
* Prior infusion reaction to a monoclonal antibody or prior hypersensitivity to Cremophor EL.
* Patients with known peripheral neuropathy (> grade 1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2004-12; Primary Completion 2007-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To determine the response rate and stable disease rate with this combination regimen

SECONDARY OUTCOMES:
To determine the clinical benefit (complete response [CR] + partial response [PR] + static disease [SD])
Time to progression
Survival rate
As well as toxicity evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Corey Langer, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Consultants in Medical Oncology & Hematology Inc., Drexel Hill, Pennsylvania, United States